CLINICAL TRIAL: NCT03468673
Title: International Validation of a Sexual Quality of Life Questionnaire Specific to HIV and Hepatitis C Infections (PROQOL-SexLife)
Brief Title: International Validation of a Sexual Quality of Life Questionnaire Specific to HIV and Hepatitis C (PROQOL-SexLife)
Acronym: SexLife
Status: Completed | Type: Observational
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: University of Sydney (Other); Center of treatment HIV/Aids-São Paulo (Unknown); Université de Montréal (Other)
Responsible Party: Principal Investigator, Dr Martin Duracinsky, Dr, University Paris 7 - Denis Diderot
Other Study IDs: PROunit PROQOL-SexLife ANRS
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Sexual Dysfunction; HIV; Hepatitis C
Keywords: AIDS; HCV; Questionnaire; Qualitative analysis; Sexual Quality of Life; Psychometric validation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop and validate a specific questionnaire of sexual quality of life in several languages and cultures (France, Brazil, Australia) allowing a meaningful and comprehensive assessment of the sexuality of patients infected with HIV and HCV; Propose reference scoring for sub-populations.

DETAILED DESCRIPTION:
Sexual health is a complex construct affecting physical, mental and social well-being. According to studies, sexual disorders are common in people with HIV infection and 25 to 71% of, both men and women regardless of their sexual orientation; and between 39 and 50 % of patients infected with Hepatitis C Virus(HCV). The cause is almost always multifactorial, with psychological, environmental and physiological components, and there may be an iatrogenic effect of treatment. HIV is a chronic disease for people with access to effective treatment. And Hepatitis C while curable is a chronic condition when untreated. In this context, sexuality is an important dimension of quality of life. But the issues are complex and not easily defined. Various studies have highlighted the lack of attention paid to sexuality in a medical management of various chronic conditions such as HIV or cancer. Indeed, a preliminary review of the literature and analysis of the concepts measured by 25 questionnaires on sexuality, shows that these instruments are inadequate to capture all aspects of the sexuality affecting quality of life of people infected with HIV or HCV. If they address physical aspects of sexuality, they address briefly at all socio-psychological and relational sexual life (body image, feeling desirable, self-esteem). Only a limited number of studies focused specifically on the experience of people suffering of sexual dysfunction in HIV and HCV infection. Moreover, these instruments do not assess specific issues related to stigma and problems related to transmission of infections of certain subgroups, particularly in the gay population.

It is an international prospective study (Australia, Brazil, Canada and France) with four phases:

Phase 1. A literature review and interview guide writing.

Phase 2. A qualitative research design based on a grounded theory research perspective:

realization and analysis of interviews with people affected by HIV and HCV, creation of the conceptual framework specific to HIV and HCV.

Phase 3. Questionnaire creation: creation of an item bank; formalization of a pilot questionnaire; forward-backward linguistic validation in each of the target languages (French, Portuguese of Brazil, English), cognitive debriefing and international harmonization; development of the conceptual model of sexual quality of life.

Phase 4. Psychometric validation of the new questionnaire: cross-sectional study by administration of the new questionnaire to 1 400 patients in the 4 countries, along with generic questionnaire about sexuality (Male sexual Health Questionnaire, Female sexual Function Index), the HIV sexual risk questionnaire, and the SF-12v2; Statistic and psychometric analysis; assessment of characteristics of different sub-populations; Propose reference scoring for sub- populations.

Impact of research: the availability of a meaningful and validated tool to detect and assess specifically sexual quality of life in HIV and HCV populations will improve the understanding of specific issues of these sub-populations. The questionnaire is intended for use in research, clinical practice, and during annual visits.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV and/or Hepatitis C
* having proficiency in English, French or Portuguese of Brazil
* Giving informed consent (oral or written consent according to the legislation of country)

Exclusion Criteria:

* cognitive impairment or major psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with HIV and / or HCV and being over the age of 18, and having proficiency in English, French or Portuguese
Sampling Method: Non-Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of a new questionnaire (PROQOL-SexLife) to assess sexual Quality of Life of people affected by HIV and HCV | 4 last weeks
  PROQOL-SexLife is the developed questionnaire through qualitative analysis (phase 2 of the study). Because it is specific to these infections, it will be used to assess the sexuality of people affected by HIV and / or Hepatitis C. This questionnaire has the potential to specifically detect sexual dysfunction. It is intended for use in research, clinical practice, and during annual visits.

CONTACTS AND LOCATIONS:
Locations (17):
- University of Sydney, Sydney, Australia
- Center of treatment HIV/Aids - Brazil, São Paulo, Brazil
- Clinique m&dicale L'Actuel, Montreal, Quebec, Canada
- France (14):
  - CHU de Bordeaux, Bordeaux
  - CHU de Dijon, Dijon
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Européen de Marseille, Marseille
  - CHU Nantes, Nantes
  - Hôpital Hôtel-Dieu, Paris
  - Hôpital Lariboisière, Paris
  - Institut Mutual Montsouris, Paris
  - Hôpital Necker, Paris
  - CHI Saint Germain en Laye, Saint-Germain-en-Laye
  - CH de Saint-Nazaire, Saint-Nazaire
  - Hôpital Foch, Suresnes
  - CHU Purpan, Toulouse
  - Centre Hépato -Biliaire de l'Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WHO | Sexual health [Internet]. WHO. Available from: http://www.who.int/topics/sexual_health/en/
- [Background] Koole O, Noestlinger C, Colebunders R. Quality of life in HIV clinical trials: why sexual health must not be ignored. PLoS Clin Trials. 2007 Mar 2;2(3):e8. doi: 10.1371/journal.pctr.0020008. No abstract available. PMID 17332849
- [Background] Marcellin F, Preau M, Ravaux I, Dellamonica P, Spire B, Carrieri MP. Self-reported fatigue and depressive symptoms as main indicators of the quality of life (QOL) of patients living with HIV and Hepatitis C: implications for clinical management and future research. HIV Clin Trials. 2007 Sep-Oct;8(5):320-7. doi: 10.1310/hct0805-320. PMID 17956833
- [Background] Sandfort TG, Collier KL, Grossberg R. Addressing sexual problems in HIV primary care: experiences from patients. Arch Sex Behav. 2013 Oct;42(7):1357-68. doi: 10.1007/s10508-012-0009-5. Epub 2012 Sep 11. PMID 22965768
- [Background] Meystre-Agustoni G, Jeannin A, de Heller K, Pecoud A, Bodenmann P, Dubois-Arber F. Talking about sexuality with the physician: are patients receiving what they wish? Swiss Med Wkly. 2011 Mar 8;141:w13178. doi: 10.4414/smw.2011.13178. eCollection 2011. PMID 21384286
- [Background] Dyer K, das Nair R. Why don't healthcare professionals talk about sex? A systematic review of recent qualitative studies conducted in the United kingdom. J Sex Med. 2013 Nov;10(11):2658-70. doi: 10.1111/j.1743-6109.2012.02856.x. Epub 2012 Jul 30. PMID 22846467
- [Background] Soykan A, Boztas H, Idilman R, Ozel ET, Tuzun AE, Ozden A, Ozden A, Kumbasar H. Sexual dysfunctions in HCV patients and its correlations with psychological and biological variables. Int J Impot Res. 2005 Mar-Apr;17(2):175-9. doi: 10.1038/sj.ijir.3901267. PMID 15510190